CLINICAL TRIAL: NCT00003562
Title: A Phase II Study of Non-Small Cell Cancer of the Lung Utilizing Low-Dose Weekly Therapy of Taxotere and Carboplatin
Brief Title: Docetaxel Plus Carboplatin in Treating Patients With Stage IIIB or Stage IV Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hope Cancer Institute, Inc. (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000066626; HCRN-007; NCI-V98-1469
Record Dates: First submitted 1999-11-01; First posted 2004-05-21 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2001-03

CONDITIONS: Lung Cancer
Keywords: squamous cell lung cancer; large cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; adenocarcinoma of the lung
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung | interventions — Carboplatin; Docetaxel

INTERVENTIONS:
Drug: carboplatin
Drug: docetaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining docetaxel and carboplatin in treating patients who have stage IIIB or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the effectiveness of low dose docetaxel and carboplatin by response rate, response duration, and time to progression in patients with stage IIIB or IV non-small cell lung cancer. II. Determine the side effects and toxicity profile of docetaxel when given in combination with carboplatin in these patients.

OUTLINE: This is open label study. Patients receive docetaxel IV over 1 hour followed by carboplatin IV over 30 minutes once a week for 4 weeks. Patients receive at least 2 courses (8 weeks) of treatment. Courses are further repeated in the absence of unacceptable toxicity and disease progression.

PROJECTED ACCRUAL: There will be 20-38 patients accrued into this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed stage IIIB with metastatic pleural effusion or metastatic stage IV non-small cell lung cancer Large cell Adenocarcinoma Squamous cell Bronchioalveolar carcinoma Undifferentiated No small cell or carcinoid histologies At least 1 bidimensionally measurable or evaluable indicator lesion Measurable or evaluable indicator lesion(s) must be completely outside the radiation portal or there must be proof of disease progression No current CNS metastases at study entry No meningeal carcinomatosis

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Zubrod 0-2 Life expectancy: Greater than 12 weeks Hematopoietic: Neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than upper limit of normal (ULN) SGOT and/or SGPT no greater than 2.5 times ULN if alkaline phosphatase less than ULN, OR alkaline phosphatase no greater than 4 times ULN if SGOT and/or SGPT less than ULN Renal: Creatinine clearance at least 50 mL/min Other: No concurrent illness that would effect assessment of this study Not pregnant or nursing Effective contraception required of all fertile patients

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior systemic chemotherapy No other concurrent chemotherapy Endocrine therapy: Not specified Radiotherapy: See Disease Characteristics Prior radiotherapy for non-small cell lung cancer allowed Radiotherapy for new brain metastases (other than leptomeningeal disease) is allowed during study, but chemotherapy is stopped during and for 2 weeks following radiotherapy Concurrent radiotherapy to other sites allowed if there is no objective criteria for disease progression Surgery: Not specified Other: No other concurrent experimental drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 1998-07

CONTACTS AND LOCATIONS:
Overall Officials: Raj Sadasivan, MD, PhD, Study Chair — Hope Cancer Institute, Inc.
Locations (2):
- United States (2):
  - Bethany Medical Center, Kansas City, Kansas
  - Heartland Cancer Research Network, Kansas City, Kansas